CLINICAL TRIAL: NCT03318133
Title: Comparison of Combined Lumbar and Sacral Plexus Block With Sedation Versus General Endotracheal Anesthesia on Postoperative Outcomes in Elderly Patients Undergoing Hip Fracture Surgery(CLSB-HIPELD): Rationale and Design of a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Comparison of CLSB With Sedation Versus General Endotracheal Anesthesia on Postoperative Outcomes in Elderly Patients Undergoing Hip Fracture Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng WANG, Attending doctor, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-28(2)
Record Dates: First submitted 2017-10-15; First posted 2017-10-23 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Anesthesia Morbidity; Anesthesia; Adverse Effect
Keywords: general anesthesia; sacral plexus block; lumbar plexus block; hip fracture; elderly
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA group (Experimental): general anesthesia(GA) group:
  1. Open peripheral vein fluid infusion, radial arterial cannulation under local lidocaine anesthesia and arterial blood pressure monitoring
  2. Propofol (1.5-3mg/kg), cis-atracurium(0.1-0.15mg/kg) and sulfentanyl(0.2-0.6μg/kg) anesthesia-induced intubation, mechanical ventilation to maintain normal PETCO2
  3. Use sevoflurane, propofol and sulfentanyl to maintain anesthesia, and add cis-atracurium as needed
  4. Transfer to ICU after surgery
  Interventions: Procedure: anesthesia
- CLSB group (Experimental): combined lumbar plexus and sacral plexus block(CLSB) group:
  1. Open peripheral vein fluid infusion
  2. In lateral position (affected side upward), ultrasound-guided lumbar plexus block (0.375% ropivacaine, Lumbar 2-3 or/and 3-4vertebral space level, 25ml), then sacral plexus block (0.375% ropivacaine, 20ml)
  3. Radial arterial cannulation under local lidocaine anesthesia and arterial blood pressure monitoring, and blockade effectiveness was evaluated 30min after nerve block
  4. After reaching satisfactory blockade, target-controlled infusion of propofol was used to maintain Ramsay sedation score between 5-6 points, monitoring PETCO2 through nasopharyngeal airway, maintain autonomous respiration, and add small-dose fentanyl (10-20μg/time) as needed
  5. Transfer to ICU after surgery
  Interventions: Procedure: anesthesia

INTERVENTIONS:
Procedure: anesthesia — in this study, we plan to make a prospective, multicenter, randomized controlled clinical trial to compare the effects of general anesthesia with endotracheal intubation and ultrasound-guided combined lumbar plexus and sacral plexus block with sedative anesthesia on the prognosis of elderly patients with hip fracture to clarify the clinical value of combined lumbar plexus and sacral plexus block with sedative anesthesia in elderly patients with hip fracture.

SUMMARY:
Hip fracture is a global public health problem. The postoperative mortality and disability rate of hip fracture is high, and early surgery is still the most effective treatment method, but these patients are often associated with concurrent heart and lung and other organ dysfunction, anesthesia and surgery are extremely risky, mainly associated with high incidence of complications in the pulmonary and cardiovascular system, and anesthesia plays a vital role in ensuring that these patients can safely and effectively get through the perioperative period.

The research on the relationship between anesthetic methods and hip fracture surgery prognosis mainly focuses on comparison between neuraxial anesthesia (including spinal anesthesia and epidural anesthesia) and general anesthesia with endotracheal intubation until now. In addition to general anesthesia with endotracheal intubation and neuraxial anesthesia, ultrasound-guided lumbar plexus and sciatic nerve block has been widely used in hip fracture surgery in recent years, especially for some high-risk patients with cardiopulmonary dysfunction. However, it is not clear whether ultrasound-guided combined lumbar plexus and sacral plexus block with sedative anesthesia can improve the prognosis of elderly patients with hip fracture, and in this study, we plan to make a prospective, multicenter, randomized controlled clinical trial to compare the effects of general anesthesia with endotracheal intubation and ultrasound-guided combined lumbar plexus and sacral plexus block with sedative anesthesia on the prognosis of elderly patients with hip fracture to clarify the clinical value of combined lumbar plexus and sacral plexus block with sedative anesthesia in elderly patients with hip fracture.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥77 years old;
2. First unilateral surgery for hip fracture including femoral neck, intertrochanteric or subtrochanteric fracture;
3. Patient with planned hip fracture surgery within 24-72 h;
4. Patient without peripheral nerve block within 24 h prior to surgery;
5. The ability to receive written informed consent from the patient or patient's legal representative.

Exclusion Criteria:

1. Refuse to participate;
2. Unable to perform nerve block;
3. Multiple trauma, multiple fractures or other fractures outside the inclusion criteria, such as pathological fractures, pelvic fractures, femur fractures;
4. Prosthetic fracture;
5. Scheduled for bilateral hip fracture surgery;
6. Usage of bone-cement fixation in the surgery;
7. With recent cerebral stroke (<3 months);
8. Combined with active heart disease (unstable angina, acute myocardial infarction, recent myocardial infarction; decompensated heart failure; symptomatic arrhythmia; severe mitral or aortic stenotic heart disease);
9. Patient with known severe lung and/or airway disease, acute respiratory failure, acute pulmonary infection, and acute attack of bronchial asthma;
10. Current enrolment in another clinical trial;
11. Contraindication for general endotracheal anesthesia(drug allergies to general anesthesia, difficult airway);
12. Contraindication for lumbar and sacral plexus block(infection at the site of needle insertion, coagulopathy, allergy to local anesthetics).

Min Age: 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1086 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality | month 1
  Telephone follow-up will be performed to confirm whether the patient survival or not after surgery.
mortality | months 3
  Telephone follow-up will be performed to confirm whether the patient survival or not after surgery.
mortality | month 6
  Telephone follow-up will be performed to confirm whether the patient survival or not after surgery.
mortality | month 12
  Telephone follow-up will be performed to confirm whether the patient survival or not after surgery.

SECONDARY OUTCOMES:
Duration of surgery | from the start to the end of the surgery
  The time spent on the surgery will be recorded.
Intraoperative complications | Intraoperative
  1. Intraoperative hypotension and vasopressor dosage
  2. Intraoperative arrhythmia, myocardial ischemia, myocardial infarction, massive hemorrhage, pulmonary embolism and hypoxemia
  3. Intraoperative blood loss and blood transfusion volume
Incidence of various complications and comprehensive complication index during hospitalization after surgery | up to 8 weeks after the surgery
SOFA score(sequential organ failure assessment score) | within 3 days after surgery
  Sepsis-related organ failure assessment score, also known as sequential organ failure assessment score (SOFA score), is used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems.Both the mean and highest SOFA scores are predictors of outcome. An increase in SOFA score during the first 24 to 48 hours in the ICU predicts a mortality rate of at least 50% up to 95%. Scores less than 9 give predictive mortality at 33% while above 11 can be close to or above 95%.
Length of stay in ICU and hospital | up to 8 weeks after the surgery
the Confusion Assessment Method(CAM) | within 3 days after surgery
  The Confusion Assessment Method includes an instrument and diagnostic algorithm for identification of delirium.The CAM instrument assesses the presence, severity, and fluctuation of 9 delirium features:acute onset, inattention, disorganized thinking, altered level of consciousness, disorientation, memory impairment, perceptual disturbances, psychomotor agitation or retardation, and altered sleep-wake cycle.
MMSE(Mini-mental State Examination) | within 3 days after surgery
  The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment. The MMSE test includes simple questions and problems in a number of areas: the time and place of the test, repeating lists of words, arithmetic such as the serial sevens, language use and comprehension, and basic motor skills.
High-sensitivity cardiac troponin T(hs-cTnT) | 1 day before surgery,1 and 3 days after surgery
  Cardiac troponin is the preferred biomarker for the diagnosis of acute myocardial infarction. A high-sensitivity cardiac troponin T(hs-cTnT) assay permits detection of very low levels of cTnT.

OTHER OUTCOMES:
Bauer Patient Satisfaction Questionnaire | on day 3 after surgery
  Satisfaction with anesthesia care will be assessed on postoperative day 3 via the Bauer Patient Satisfaction Questionnaire. The questionnaire enables a consistent, reliable and valid evalution of patient satisfaction with anesthesia care.
Economic parameters | on day 1 after discharge
  Economic parameters including total cost in hospital and expenditure for anesthesia
Barthel Activities of Daily Living Index | on day 30 after discharge and surgery
  Functional recovery on day 30 after discharge and surgery, evaluated by Barthel Activities of Daily Living Index. Assesses functional independence, generally in stroke patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang J, Wang X, Zhang H, Shu Z, Jiang W. Comparison of combined lumbar and sacral plexus block with sedation versus general anaesthesia on postoperative outcomes in elderly patients undergoing hip fracture surgery (CLSB-HIPELD): study protocol for a prospective, multicentre, randomised controlled trial. BMJ Open. 2019 Mar 30;9(3):e022898. doi: 10.1136/bmjopen-2018-022898. PMID 30928924